CLINICAL TRIAL: NCT04247126
Title: A Phase 1 Study of SY 5609, an Oral, Selective CDK7 Inhibitor, in Adult Patients With Select Advanced Solid Tumors
Brief Title: A Study of SY 5609, a Selective CDK7 Inhibitor, in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syros Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SY-5609-101
Record Dates: First submitted 2020-01-22; First posted 2020-01-29 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor; Breast Cancer; Small-cell Lung Cancer; Pancreatic Cancer
MeSH Terms: conditions — Breast Neoplasms; Small Cell Lung Carcinoma; Pancreatic Neoplasms | interventions — SY-5609; Fulvestrant; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Single Agent Dose Escalation (Experimental): Dose escalation phase to explore maximum tolerated dose of SY-5609 given as a single agent.
  Interventions: Drug: SY-5609
- Group 2: SY-5609 + Fulvestrant (Experimental): Participants with hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2) negative advanced or metastatic breast cancer (BC) that has progressed following prior treatment with a cyclin-dependent kinase (CDK)4/6 inhibitor in combination with hormonal therapy will receive SY-5609 in combination with fulvestrant.
  Interventions: Drug: SY-5609; Drug: Fulvestrant
- Group 3: SY-5609 + Gemcitabine (Experimental): Participants with PDAC will receive SY-5609 in combination with gemcitabine in Safety Lead-in to identify a recommended combination dose for the expansion. The expansion part will assess the safety, tolerability, and preliminary clinical activity of SY-5609 in combination with gemcitabine at the recommended combination dose.
  Interventions: Drug: SY-5609; Drug: Gemcitabine
- Group 4: SY-5609 + Gemcitabine + Nab-paclitaxel (Experimental): Participants with PDAC will receive SY-5609 in combination with gemcitabine plus nab-paclitaxel in Safety Lead-in to identify a recommended combination dose for the expansion. The expansion part will assess the safety, tolerability, and preliminary clinical activity of SY-5609 in combination with gemcitabine plus nab-paclitaxel at the recommended combination dose.
  Interventions: Drug: SY-5609; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: SY-5609 — An oral CDK7 Inhibitor
Drug: Fulvestrant — Estrogen receptor antagonist
  Arms: Group 2: SY-5609 + Fulvestrant
Drug: Gemcitabine — Nucleoside metabolic inhibitor
  Arms: Group 3: SY-5609 + Gemcitabine; Group 4: SY-5609 + Gemcitabine + Nab-paclitaxel
Drug: Nab-paclitaxel — Taxane-type chemotherapy
  Arms: Group 4: SY-5609 + Gemcitabine + Nab-paclitaxel

SUMMARY:
The study consists of 2 parts. Part 1 is dose escalation and will first administer SY-5609 alone to participants with select advanced solid tumors and then in combination with fulvestrant to participants with HR positive, HER2-negative breast cancer. Part 2 is a dose expansion and will first administer SY-5609 in combination with gemcitabine and then SY-5609 in combination with gemcitabine and nab-paclitaxel in participants with pancreatic ductal adenocarcinoma (PDAC) .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Advanced Solid Tumors for which standard curative or palliative measures do not exist or are no longer effective (Group 1 only).
3. Postmenopausal women with HR-positive, HER2-negative advanced or metastatic breast cancer. Participants must have failed prior treatment with a cyclin-dependent kinase (CDK) 4/6 inhibitor in combination with hormonal therapy in a previous line of therapy (Group 2 only).
4. Participants with histologically or cytologically confirmed PDAC with measurable metastatic lesion(s) (Groups 3 and 4 only).
5. Participants must have at least 1 measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
6. All toxicities (except alopecia) from prior cancer treatments must have resolved to ≤ Grade 1 before enrollment.
7. For women of childbearing potential (WCBP): negative serum β human chorionic gonadotropin pregnancy test within 1 week before the first dose of SY 5609
8. Adequate organ and marrow function
9. Participants must be willing and able to comply with all aspects of the protocol
10. Participants must provide written informed consent before any study-specific screening procedures.
11. Albumin ≥ 3.0 grams/deciliters (g/dL) (Groups 3 and 4 only).

Exclusion Criteria:

1. Chemotherapy or limited field radiotherapy within 2 weeks, wide field radiotherapy within 4 weeks, or nitrosoureas or mitomycin C within 6 weeks before entering the study
2. Major surgery within 2 weeks before starting the study treatment, or not recovered to baseline status from the effects of surgery received > 2 weeks prior
3. Received any other investigational agents within 4 weeks before enrollment, or < 5 half-lives since completion of previous investigational therapy, whichever is shorter
4. Received previous noncytotoxic, US Food and Drug Administration-approved anticancer agent within previous 2 weeks, or < 5 half-lives since completion of previous therapy, whichever is shorter
5. Known brain metastases or carcinomatous meningitis
6. Immunocompromised participants with increased risk of opportunistic infections
7. Participants with known active or chronic hepatitis B or active hepatitis C infection. Participants with a history of hepatitis C virus (HCV) infection who have completed curative therapy for HCV at least 12 weeks before Screening and have a documented undetectable viral load at Screening are eligible for enrollment.
8. Baseline QT interval corrected (QTc) with Fridericia's method > 480 milliseconds

   • NOTE: criterion does not apply to participants with a right or left bundle branch block (QTc interval)
9. Female participants who are pregnant or breastfeeding
10. History of clinically significant cardiac disease or clinically relevant uncontrolled cardiac risk factors
11. Uncontrolled intercurrent illness.
12. Poorly controlled ascites requiring paracentesis within 1 month prior to entering the study. (Groups 3 and 4 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Groups 1 and 2: Dose-Limiting Toxicity of SY-5609 | Up to 28 days after first administration
Groups 1 and 2: Number of Participants With Treatment Emergent Adverse Events | From Baseline up to 30 days after last dose of study drug (up to 1 year)
Groups 3 and 4 (Safety Lead-ins): Number of Participants With Dose-Limiting Toxicity | Up to 28 days after first administration
Groups 3 and 4 (Safety Lead-ins): Number of Participants With TEAEs | From Baseline up to 30 days after last dose of study drug (up to 1 year)
Groups 3 and 4 (Expansions): Progression Free Survival | Up to 1 year

SECONDARY OUTCOMES:
Groups 1 and 2: Area Under The Concentration Versus Time Curve of SY-6509 | Predose, 0.5, 1, 2, 4, 6, 8 hours postdose on Day 1 and 4 or 15 of Cycle 1; 24 hours predose on Day 2 and 5 of Cycle 1; 24 hours predose on Day 1 of Cycle 2, 3 and 4 (Each Cycle=28 days)
Groups 1 and 2: Apparent Clearance of SY-5609 | Predose, 0.5, 1, 2, 4, 6, 8 hours postdose on Day 1 and 4 or 15 of Cycle 1; 24 hours predose on Day 2 and 5 of Cycle 1; 24 hours predose on Day 1 of Cycle 2, 3 and 4 (Each Cycle=28 days)
Groups 1 and 2: Apparent Volume of Distribution of SY-5609 | Predose, 0.5, 1, 2, 4, 6, 8 hours postdose on Day 1 and 4 or 15 of Cycle 1; 24 hours predose on Day 2 and 5 of Cycle 1; 24 hours predose on Day 1 of Cycle 2, 3 and 4 (Each Cycle=28 days)
Groups 1 and 2: Elimination Half-Life of SY-5609 | Predose, 0.5, 1, 2, 4, 6, 8 hours postdose on Day 1 and 4 or 15 of Cycle 1; 24 hours predose on Day 2 and 5 of Cycle 1; 24 hours predose on Day 1 of Cycle 2, 3 and 4 (Each Cycle=28 days)
Groups 1 and 2: Maximum Plasma Concentration (Cmax) of SY-5609 | Predose, 0.5, 1, 2, 4, 6, 8 hours postdose on Day 1 and 4 or 15 of Cycle 1; 24 hours predose on Day 2 and 5 of Cycle 1; 24 hours predose on Day 1 of Cycle 2, 3 and 4 (Each Cycle=28 days)
Groups 1 and 2: Time of Maximum Plasma Concentration (Tmax) of SY-5609 | Predose, 0.5, 1, 2, 4, 6, 8 hours postdose on Day 1 and 4 or 15 of Cycle 1; 24 hours predose on Day 2 and 5 of Cycle 1; 24 hours predose on Day 1 of Cycle 2, 3 and 4 (Each Cycle=28 days)
Groups 1 and 2: Minimum or Trough Plasma Concentration (Cmin) of SY-5609 | Predose, 0.5, 1, 2, 4, 6, 8 hours postdose on Day 1 and 4 or 15 of Cycle 1; 24 hours predose on Day 2 and 5 of Cycle 1; 24 hours predose on Day 1 of Cycle 2, 3 and 4 (Each Cycle=28 days)
Groups 1 and 2: Time of Minimum or Trough Plasma Concentration (Tmin) of SY-5609 | Predose, 0.5, 1, 2, 4, 6, 8 hours postdose on Day 1 and 4 or 15 of Cycle 1; 24 hours predose on Day 2 and 5 of Cycle 1; 24 hours predose on Day 1 of Cycle 2, 3 and 4 (Each Cycle=28 days)
Groups 3 and 4 (Safety Lead-ins): Progression Free Survival | Up to 1 year
Groups 3 and 4 (Safety Lead-ins): Objective Response Rate (ORR) | Up to 1 year
  ORR is defined as the proportion of participants who achieve complete response (CR) and partial remission (PR) (as determined by the investigator).
Groups 3 and 4 (Safety Lead-ins): Complete Response/Remission (CR) Rate | Up to 1 year
  CR rate is defined as proportion of participants who achieve CR (as determined by the investigator).
Groups 3 and 4 (Safety Lead-ins): Disease Control Rate | Up to 1 year
Groups 3 and 4 (Safety Lead-ins): Time to Response | Up to 1 year
  Time to response is defined as the duration from the date of randomization to the date of the first documented evidence of response as determined by the investigator.
Groups 3 and 4 (Safety Lead-ins): Duration of Response | Up to 1 year
  Duration of response is defined as duration from the date of first documented evidence of response to the date of relapse of disease (as determined by the investigator), or death due to any cause, whichever occurs first.
Groups 3 and 4 (Expansions): Objective Response Rate | Up to 1 year
  ORR is defined as the proportion of participants who achieve CR and partial remission (PR) (as determined by the investigator).
Groups 3 and 4 (Expansions): Complete Response Rate | Up to 1 year
  CR rate is defined as proportion of participants who achieve CR (as determined by the investigator).
Groups 3 and 4 (Expansions): Disease Control Rate | Up to 1 year
Groups 3 and 4 (Expansions): Time to Response | Up to 1 year
  Time to response is defined as the duration from the date of randomization to the date of the first documented evidence of response as determined by the investigator.
Groups 3 and 4 (Expansions): Duration of Response | Up to 1 year
  Duration of response is defined as duration from the date of first documented evidence of response to the date of relapse of disease (as determined by the investigator), or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Orlando Health Cancer Institute, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - The University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - START Midwest, LLC, Grand Rapids, Michigan
  - Duke University, Durham, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - South Texas Accelerated Research Theraputics (START), LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marineau JJ, Hamman KB, Hu S, Alnemy S, Mihalich J, Kabro A, Whitmore KM, Winter DK, Roy S, Ciblat S, Ke N, Savinainen A, Wilsily A, Malojcic G, Zahler R, Schmidt D, Bradley MJ, Waters NJ, Chuaqui C. Discovery of SY-5609: A Selective, Noncovalent Inhibitor of CDK7. J Med Chem. 2022 Jan 27;65(2):1458-1480. doi: 10.1021/acs.jmedchem.1c01171. Epub 2021 Nov 2. PMID 34726887
- [Derived] Sava GP, Fan H, Coombes RC, Buluwela L, Ali S. CDK7 inhibitors as anticancer drugs. Cancer Metastasis Rev. 2020 Sep;39(3):805-823. doi: 10.1007/s10555-020-09885-8. PMID 32385714